CLINICAL TRIAL: NCT01447472
Title: Human Study of the Metabolic Changes Induced by 3,4-methylenedioxymethamphetamine (MDMA, Ecstasy) in the Metabolism of Dextromethorphan and Caffeine
Brief Title: -Methylenedioxymethamphetamine (MDMA, Ecstasy) Induced Changes in Drug Metabolism: Gender and Genetic Polymorphisms
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: IMIMFTCL/MDMA/6; AEMPS no.04-0013 (Other: Spanish Medicines Agency (identification number)); 5R01DA017987 (NIH)
Record Dates: First submitted 2011-09-27; First posted 2011-10-06 (Estimated); Last update posted 2011-10-06 (Estimated); Status verified 2011-10

CONDITIONS: Metabolism; Interaction
Keywords: MDMA,; pharmacokinetics,; pharmacodynamics,; CYP2D6, COMT,; SERT, 5-HTTLPR, gender,; dextromethorphan,; caffeine.
MeSH Terms: conditions — Coitus | interventions — N-Methyl-3,4-methylenedioxyamphetamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MDMA (Experimental): One single dose of MDMA (1.5 mg/kg; range 75-100 mg)
  Interventions: Drug: MDMA

INTERVENTIONS:
Drug: MDMA — One single dose of MDMA ( 1.5 mg/kg; range: 75-100 mg)
  Other Names: Ecstasy

SUMMARY:
The purpose of this study are:

1. to evaluate the involvement of CYP2D6, CYP3A4 and CYP1A2 (through dextromethorphan and caffeine challenges), and catechol-O-methyltransferase (COMT)in MDMA metabolism
2. to evaluate gender differences in the human pharmacology of MDMA
3. to study the influence of some genetic polymorphisms (CYP2D6, COMT, SERT) in the effects and pharmacokinetics of MDMA.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female adults, the recreational use of MDMA on at least ten occasions (two in the previous year), and the EM phenotype for CYP2D6 activity determined using dextromethorphan as a selective probe drug.
* Women had to present a regular menstrual cycle and not take oral contraceptives.

Exclusion Criteria:

* Daily consumption >20 cigarettes and >4 standard units of ethanol in men (>2 in women)
* Regular ingestion of medication in the month preceding the study
* Presence of major psychiatric disorders
* History of abuse or drug dependence (except for nicotine dependence)
* Psychiatric adverse reactions after MDMA consumption.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2003-05; Primary Completion 2009-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Concentrations of dextromethorphan in plasma and urine. | 240 hours after MDMA dosing.
  Blood samples and urine to determine dextromethorphan and dextrorphan concentrations until 240h.
Concentrations of caffeine in plasma and urine. | 24 hours after MDMA dosing.
  Blood samples and urine to determine caffeine and theobromine concentrations until 240h.
Concentrations of MDMA and metabolites (influence of gender) | 48h after MDMA administration.
  Determination of MDMA and metabolites concentrations in plasma and urine during 48h. Influence of gender male/female.
Concentrations of MDMA and metabolites (influence of genetics) | 48h after MDMA administration.
  Determination of MDMA and metabolites concentrations in plasma and urine during 48h. Influence of gene polymorphisms of CYP2D6, CYP3A4, COMT, SERT.

SECONDARY OUTCOMES:
Effects of MDMA on physiological response. | 24h
  Effects of MDMA on blood preassure, heart rate, temperature, pupil diameter, esophoria. Influence of gender and genetic polymorphisms.
Effects of MDMA on physiological response. | 24h
  Effects of MDMA on subjective effects (feelings of intoxication, euphoria, bad effects etc) and psychological tests (VESSPA, ARCI). Influence of gender and genetic polymorphisms.

CONTACTS AND LOCATIONS:
Overall Officials: Magí Farre, PhD, Principal Investigator — IMIM-Hospital del Mar (Institut de Recerca Hospital del Mar)
Locations (1):
- IMIM-Hospital del Mar (Institut de Recerca Hospital del Mar), Barcelona, Barcelona, Spain

REFERENCES:
- [Result] Yubero-Lahoz S, Pardo R, Farre M, O'Mahony B, Torrens M, Mustata C, Perez-Mana C, Carbo ML, de la Torre R. Sex differences in 3,4-methylenedioxymethamphetamine (MDMA; ecstasy)-induced cytochrome P450 2D6 inhibition in humans. Clin Pharmacokinet. 2011 May;50(5):319-29. doi: 10.2165/11584550-000000000-00000. PMID 21456632
- [Result] O'Mathuna B, Farre M, Rostami-Hodjegan A, Yang J, Cuyas E, Torrens M, Pardo R, Abanades S, Maluf S, Tucker GT, de la Torre R. The consequences of 3,4-methylenedioxymethamphetamine induced CYP2D6 inhibition in humans. J Clin Psychopharmacol. 2008 Oct;28(5):523-9. doi: 10.1097/JCP.0b013e318184ff6e. PMID 18794647
- [Derived] Pardo-Lozano R, Farre M, Yubero-Lahoz S, O'Mathuna B, Torrens M, Mustata C, Perez-Mana C, Langohr K, Cuyas E, Carbo Ml, de la Torre R. Clinical pharmacology of 3,4-methylenedioxymethamphetamine (MDMA, "ecstasy"): the influence of gender and genetics (CYP2D6, COMT, 5-HTT). PLoS One. 2012;7(10):e47599. doi: 10.1371/journal.pone.0047599. Epub 2012 Oct 24. PMID 23112822